CLINICAL TRIAL: NCT04639856
Title: ICU Stay in Patients With Low Ejection Fraction Undergoing Cardiac Revascularization: Comparison of On-pump vs Off-pump Coronary Artery Bypass Grafting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Armed Forces Institute of Cardiology, Pakistan (Other)
Responsible Party: Principal Investigator, Muhammad Bilal, Cardiac Surgeon, Armed Forces Institute of Cardiology, Pakistan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AFIC-IERB-SOP-15
Record Dates: First submitted 2020-11-17; First posted 2020-11-23 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: Cardiac Revascularization
Keywords: Coronary Artery Bypass Grafting
MeSH Terms: interventions — Coronary Artery Bypass

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- on-pump CABG (Active Comparator): CABG using Cardiopulmonary Bypass Machine
  Interventions: Procedure: Coronary Artery Bypass Grafting
- off-pump CABG (Active Comparator): CABG without Cardiopulmonary Bypass Machine
  Interventions: Procedure: Coronary Artery Bypass Grafting

INTERVENTIONS:
Procedure: Coronary Artery Bypass Grafting — on-pump vs off pump Coronary artery Bypass Grafting

SUMMARY:
Coronary artery bypass graft (CABG) surgery can result in severe postoperative complications, such as renal and pulmonary failure. In about 80% of the cases worldwide, it is currently performed with cardiopulmonary bypass (CPB) with cardiac arrest. Cardiopulmonary bypass leads to a systemic inflammatory response, which may be induced by the contact of circulating blood with artificial surfaces of the extracorporeal circuit.[1] To reduce postoperative complications caused by systemic inflammation, off-pump CABG was reintroduced into clinical practice in the early 1990s. During off-pump surgery, the coronary artery grafts are placed on coronaries of a beating heart, thereby avoiding aortic cross clamping and CPB. [1] There are many studies and debates about the two approaches to cardiac revascularization via CABG. This study aims to answer the question as to difference in the ICU stay of patients with low ejection fraction undergoing cardiac revascularization bet ween off pump and on pump coronary artery bypass grafting and better treatment option shall be adopted in future.

ELIGIBILITY:
Inclusion Criteria:

* All patients of either gender between the ages of 40 to 80
* Ejection fraction of less than or equal to 35% undergoing CABG.
* undergoing CABG.

Exclusion Criteria:

* Patients with ejection fraction of more than 35%
* Patients with previous history of cardiac revascularization
* Patients with previous history of chronic kidney disease and obstructive sleep apnea.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2018-07-15 (Actual); Primary Completion 2019-01-15 (Actual); Study Completion 2019-01-15 (Actual)

PRIMARY OUTCOMES:
ICU Stay | 6 Months
  post operative ICU stay in patients undergoing cardiac revascularization

CONTACTS AND LOCATIONS:
Locations (1):
- Armed Forces Institute of Cardiology, Rawalpindi, Rawalpindi, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP